CLINICAL TRIAL: NCT07300137
Title: Comparison of Outcome of Amniotic Membrane Dressing vs Sodium Carboxylic Methyl Cellulose Silver Dressing (Aquacel®Ag) in Terms of Healing in Second-Degree Burns - A Randomized Controlled Trial''
Brief Title: Comparison of Amniotic Membrane Dressing and Aquacel®Ag in Second-degree Burns
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Patel Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Shazra Khalid, Resident Plastic Surgery, Patel Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RFC_024
Record Dates: First submitted 2025-12-03; First posted 2025-12-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Second Degree Burns
Keywords: second degree burns.; amniotic membrane.; Aqua cel.; wound healing.

STUDY DESIGN:
Masking Description: analyst only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amniotic membrane dressing group (Experimental): application of preserved amniotic membrane dressing on second degree burns until healed
  Interventions: Biological: preserved amniotic membrane dressing
- Aqua cel (Ag) dressing group (Active Comparator): application of aqua cel dressing on second degree burns until healed
  Interventions: Biological: preserved amniotic membrane dressing

INTERVENTIONS:
Biological: preserved amniotic membrane dressing — application of preserved human amniotic membrane as a biological dressing for second degree burn wounds

SUMMARY:
To compare the outcome of amniotic membrane dressing versus Aquacel® Ag dressing with respect to the duration of healing in patients with second-degree burns within the local demographic setting. This study aims to address the existing gap in the literature by comparing the efficacy of amniotic membrane dressing and Aquacel® Ag dressing in the management of second-degree burns. Although Aquacel® Ag has been extensively studied for partial-thickness burns, it has not been directly compared with human amniotic membrane dressing, and no randomized controlled trial has yet evaluated these two treatment modalities. The findings of this study are expected to provide healthcare providers with an effective and cost-efficient dressing option for burn patients, particularly in resource-limited countries, while minimizing morbidity.

DETAILED DESCRIPTION:
Burns pose a significant global health burden, particularly in low- and middle-income countries. Optimal wound care is essential to enhance healing, reduce complications, and minimize the need for surgical interventions. Human amniotic membrane dressings and silver-impregnated hydrofiber dressings such as Aquacel® Ag are commonly used options for the management of second-degree burns, each offering distinct biological properties and clinical benefits.

This randomized controlled trial aims to compare the efficacy of amniotic membrane dressing with Aquacel® Ag (sodium carboxymethylcellulose silver dressing) in terms of wound healing in patients with second-degree burns. The study will include patients presenting within 72 hours of injury with burns involving ≤40% total body surface area (TBSA). A total of 100 participants will be enrolled using non-probability convenience sampling and randomized through a computer-generated method into two groups. Group A will receive amniotic membrane dressings, while Group B will be treated with Aquacel® Ag dressings.

In Group A, dressings will be changed every 72 hours. In Group B, secondary dressings will be changed and the wound will be reviewed for soakage or gross contamination, with dressings continued until complete wound healing is achieved. Based on the study hypothesis, amniotic membrane dressings are expected to provide a clinically superior alternative to Aquacel® Ag dressings in the management of second-degree burns, particularly with respect to healing time and participant comfort.

ELIGIBILITY:
Inclusion Criteria:

* second degree burns (till 40% TBSA)
* In patients/ OPD
* Fire Burn, Scald Burn, Flash Burn.

Exclusion Criteria:

* Referred Cases, Infected Wounds, Diabetic Patients/ on immunosuppressants/ corticosteroids,
* Electrical & Chemical Burns/

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Healing | 21days
  comparison of healing time between aqua cel and amniotic membrane dressing

CONTACTS AND LOCATIONS:
Overall Officials: Shazra Khalid, MBBS, Principal Investigator — Patel Hospital
Locations (1):
- Patel hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
IPD as per performa / questionnaire will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: When study will be published
Access Criteria: anyone who asks for it
URL: http://example.com

REFERENCES:
- See also: Published article providing background information on the comparison of sodium carboxylic methyl-cellulose silver dressing versus standard petroleum gauze dressing for management of second-degree burns. — https://pjmhsonline.com/index.php/pjmhs/article/view/3992
- Available data/document: comparison between two types of dressings: comparison of 2 dressings — https://pjmhsonline.com/index.php/pjmhs/article/view/3992 — Mean duration of healing with sodium Carboxylic methyl-cellulose silver dressing was less than petroleum gauze dressing for management of second-degree burns.